CLINICAL TRIAL: NCT06512103
Title: Relationship Between Bone Resorption and Sclerostin Regulation in Apical Periodontitis Lesions
Brief Title: Sclerostin Regulation in Apical Periodontitis Lesions in Apical Periodontitis Lesions
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Seyda Ersahan, DDS, PhD, Principal Investigator, Clinical Associate Professor, Istanbul Medipol University Hospital
Other Study IDs: 623
Record Dates: First submitted 2024-05-16; First posted 2024-07-22 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-07

CONDITIONS: Apical Periodontitis
Keywords: Apical periodontitis; Bone resorption; Gingival crevicular fluid; Sklerostin; PGE2
MeSH Terms: conditions — Periapical Periodontitis; Bone Resorption

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental: 90 patients with apical periodontitis (AP group): AP group was divided into 3 subgroups. The participants in the study group were divided into two subgroups: 35 patients with a PAI score of 3-4 (Group 2: mild-moderate AP), and 55 patients with at least one tooth with a severity of PAI 5 (Group 3: Severe AP).
  Interventions: Diagnostic Test: Apical periodontitis group
- Control: A healthy control group of 35 volunteers: A healthy control group of 35 volunteers without periodontal pathology as well as any acute/chronic disease (muscle-joint-bone diseases, inflammatory bowel disease, local or generalized infection, severe organ disease, cardiovascular disease and diabetes mellitus), were included in the control group. 35 healthy patients with a PAI score of 1-2 (Group 1: Control group) were included.
  Interventions: Diagnostic Test: Apical periodontitis group

INTERVENTIONS:
Diagnostic Test: Apical periodontitis group — Radiography of the patients were taken. Blood samples and gingival crevicular fluid samples were collected from those patient
  Other Names: Control group

SUMMARY:
Our aim was to examine the relationship between inflammatory bone resorption associated with the severity of AP and gingival crevicular fluid (GCF) and blood sclerostin and PGE2 levels in cases of AP. Additionally, the correlation of sclerostin regulation with RANKL and MMP-9 levels will be investigated.This single-centered cross-sectional analytical study included 90 patients with AP and 35 systemically and orally healthy volunteers as the control group, who applied for a control examination between September 2023 and February 2024. Demographic characteristics of the patients (age, body mass index (BMI) and oral hygiene index (OHI)) and dental examination findings (periapical index (PAI) score, root canal treatment, number of crowns, fillings and missing teeth, etc.) were recorded. According to the PAI score, the participants were divided into three groups: 35 healthy patients with a PAI score of 1-2 (Group 1: Control group), 35 patients with a PAI score of 3-4 (Group 2: mild-moderate AP), and 55 patients having at least one tooth with PAI score of 5, characterized by more severe bone resorption (Group 3: Severe AP). Sclerostin, RANKL and MMP-9 levels were measured in serum and GCF of all participants.

DETAILED DESCRIPTION:
Fasting (8-10 hours) venous blood of all participants was taken from forearm antecubital/basic veins. After keeping the blood at room temperature for 30 minutes, it was centrifuged at 2500 xg for 10 minutes. After centrifugation, the upper serum of the tubes was separated. Hemolysis index (HI) of the sera were measured to prevent optical interference in the biochemistry autoanalyzer device (Cobas 8000 Chemistry Analyzer, USA). Samples with a hemolysis index greater than 50 mg/dl Hb were excluded from the study. The sera obtained after centrifugation were aliquoted into 0.5 mL tubes (Eppendorf, Hamburg, Germany) and stored at - 80 °C until the day of analysis.

GCF samples were taken prior to periodontal probing to avoid contamination by blood. To avoid contamination of the sample, patients were asked not to eat or drink anything for at least 30 minutes before the procedure. After selecting the area where GCF collection would be made (the area of the tooth with AP and the area that often corresponds to the same area in healthy individuals), the sampling area was isolated with cotton rolls, and plaque was removed. After gentle air-drying, PerioPaper strips (OraFlow Inc., NY, USA) were placed gently until slight resistance was felt and left there for 30 seconds. Three samples were taken from the mesial, distal and buccal surfaces of related tooth. Periopapers were thoroughly washed in 0.5 ml Eppendorf tubes (after subtracting the tare weight of the tube) with 100 µl of phosphate-buffered saline (PBS) using an automatic pipette. Blood-stained paper strips were removed from the samples. All GCF samples were weighed on a precision balance (Shimadzu Libror, Model AEG-220, Germany) and recorded. The samples in all closed tubes were mixed thoroughly with a vortex device (Heidolph Reax Top Vortex, Schwabach, Germany) for approximately 15-20 seconds. This allowed GCF to pass into PBS. Periopapers in tubes were removed from GCF and PBS without contamination. The remaining extract in tubes was stored at -80oC until the day of analysis. The results obtained on the study day were proportioned by weighing weights/PBS. On the day of analysis, all serums and GCF were first allowed to dissolve slowly at +4 oC and then brought to room temperature before measurement.

ELIGIBILITY:
Inclusion Criteria:

patients with chronic apical periodontitis having no periodontal pathology having no acute/chronic disease (muscle-joint-bone diseases, inflammatory bowel disease, local or generalized infection, severe organ disease, cardiovascular disease and diabetes mellitus)

Exclusion Criteria:

Patients who had any acute/chronic disease (inflammatory and rheumatoid diseases, cardiovascular disease, muscle-joint-bone diseases, inflammatory bowel disease, local or generalized infection, connective tissue diseases and diabetes mellitus) patients who had a history of smoking pregnant and/or lactating patients antibiotics or anti-inflammatory drugs use within the last 6 months patients undergoing dental treatment having chronic marginal periodontitis along with AP patients with a history of using immunosuppressive drugs, steroid or nonsteroidal anti-inflammatory drugs use of high doses of biotin vitamin in the last 48 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included 90 patients diagnosed with chronic apical periodontitis. 35 healthy volunteers who came to the dental clinic for check-up and periodic examination and did not have periodontal pathology, any acute/chronic disease.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
levels of sclerostin, RANKL, MMP-9 and PGE2 in gingival crevicular fluid | baseline
  correlation between periapical radiolucency and GCF levels will be evaluated

SECONDARY OUTCOMES:
levels of sclerostin, RANKL, MMP-9 and PGE2 in serum | baseline
  correlation between periapical radiolucency and serum levels will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Uysal, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Upon request from corresponding author, we can share our data